CLINICAL TRIAL: NCT03783338
Title: Interaction Effects of Vitamin D Supplementation and Aerobic Exercises on Balance and Physical Performance in Children With Down Syndrome
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Mohamed Ahmed Mahmoud Eid, Assistant Professor, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: P.T.REC/012/002143
Record Dates: First submitted 2018-12-17; First posted 2018-12-21 (Actual); Last update posted 2019-12-02 (Actual); Status verified 2019-11

CONDITIONS: Children With Down Syndrome
Keywords: Aerobic exercises; Balance; Down syndrome; Physical performance; Vitamin D
MeSH Terms: conditions — Down Syndrome | interventions — Exercise

STUDY DESIGN:
Intervention Model Description: Children will be assigned randomly using sealed envelopes into three intervention groups (A, B and C groups). Group A will receive the conventional physical therapy program (CPTP) only. Group B will receive the CPTP in addition to aerobic exercises, whereas group C will receive CPTP, aerobic exercises in addition to an oral daily dose of vitamin D3 1000 IU (Cholecalciferol). All groups will receive the treatment program for 12 weeks.
Who Masked: Outcomes Assessor
Masking Description: The outcomes assessor will be blinded to which each child allocated to any one of the three arms.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Physical therapy group (Active Comparator): Group A will consist of 15 children and will receive the conventional physical therapy program only. This group will be used to compare the results of the other two groups.
  Interventions: Combination Product: Aerobic exercises and Vitamin D supplementation
- Physical therapy and aerobic exercises group (Experimental): Group B will consist of 15 children and will receive the conventional physical therapy program and aerobic exercises.
  Interventions: Combination Product: Aerobic exercises and Vitamin D supplementation
- Physical therapy, aerobic exercises and vitamin D group (Experimental): Group C will consist of 15 children and will receive the conventional physical therapy program, aerobic exercises and an oral daily dose of vitamin D3 1000 IU (Cholecalciferol) .
  Interventions: Combination Product: Aerobic exercises and Vitamin D supplementation

INTERVENTIONS:
Combination Product: Aerobic exercises and Vitamin D supplementation — Aerobic exercises:
  Children in groups B and C will receive aerobic exercises in the form of bicycle ergometer and treadmill training for 15 min 3 days/week for 12 weeks. The procedure and goals of exercise will be explained to all children before starting the exercise program. The child will stop exercising immediately if he feels pain, fainting or shortness of breath.
  Vitamin D supplementation:
  Children in group C only will receive vitamin D supplementation in the form of an oral daily dose of vitamin D3 1000 IU (Cholecalciferol) for 12 weeks.

SUMMARY:
Objective: To investigate the interaction effects of vitamin D supplementation and aerobic exercises on balance control and physical performance in children with Down syndrome (DS).

Methods: Forty-five children with DS ranging in age from 8 to 12 years will be selected and will participate in this study. They will be assigned randomly using sealed envelopes into three equal groups (A, B and C). Group A will consist of 15 children and will receive the conventional physical therapy program (CPTP) only. Group B will consist of 15 children and will receive the CPTP plus the aerobic exercises. Group C also will consist of 15 children and will receive the CPTP, the aerobic exercises and Vitamin D supplementation in the form of an oral dose of vitamin D3 1000 IU (Cholecalciferol). The program of treatment will be 3 days/week for 12 weeks. Evaluation of balance by using the biodex balance system and physical performance by using the six-minute walk test (6MWT) will be conducted at baseline and after 12 weeks of the treatment program.

ELIGIBILITY:
Inclusion Criteria:

* Children with DS who can stand and walk independently
* Children with 25 (OH) vitamin D levels of 16 ng/ml or less
* Children who are not consuming estrogens, steroids or other medications that could interfere with vitamin D metabolism
* The absence of visual and hearing impairments that could interfere with testing and training protocols
* Children with mild intellectual disabilities and were capable of understanding visual and verbal instructions.

Exclusion Criteria:

* Medical conditions that will severely limit a child's participation in the study as cardiac problems.
* Musculoskeletal deformities of the lower limbs.

Ages: 8 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 59 (Actual)
Dates: Start 2018-12-02 (Actual); Primary Completion 2019-03-02 (Actual); Study Completion 2019-03-02 (Actual)

PRIMARY OUTCOMES:
Balance | This outcome will be measured for each child before the beginning of treatment program and immediately after 12 weeks of the treatment program.
  Balance assessment will be conducted by using the Biodex Stability System (BSS; Biodex, Inc, Shirley, NY) that enables objective assessment of balance.
Physical performance | This outcome will be measured for each child before the beginning of treatment program and immediately after 12 weeks of the treatment program.
  Physical performance will be evaluated using the six-minute walk test (6MWT).

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty of Physical Therapy - Cairo University, Cairo, Giza Governorate, Egypt

IPD SHARING:
Plan to Share IPD: Undecided